CLINICAL TRIAL: NCT04743154
Title: In-hospital Versus After-discharge Complete Revascularization in STEMI Patients With Multivessel Disease.
Brief Title: In-hospital Versus After-discharge Complete Revascularization
Acronym: REVIVA-ST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital General Universitario de Valencia (Other)
Responsible Party: Principal Investigator, Eva Rumiz González, Principal investigator, Hospital General Universitario de Valencia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: HGUValencia
Record Dates: First submitted 2021-02-03; First posted 2021-02-08 (Actual); Last update posted 2023-04-24 (Actual); Status verified 2023-04

CONDITIONS: STEMI - ST Elevation Myocardial Infarction; Multivessel Coronary Artery Disease
Keywords: STEMI; Multivessel; PCI
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- In-hospital complete revascularization group. (Other): Patients will undergo to a complete revascularization of non-culprit lesions at least 24 hours after STEMI and before hospital discharge.
  Interventions: Other: In-hospital nonculprit-lesions percutaneous coronary intervention (PCI)
- After-discharge complete revascularization group. (Other): Patients will undergo to a complete revascularization of non-culprit lesions after hospital discharge within 4-6 weeks after STEMI.
  Interventions: Other: After-discharge nonculprit-lesions percutaneous coronary intervention (PCI)

INTERVENTIONS:
Other: In-hospital nonculprit-lesions percutaneous coronary intervention (PCI) — To perform percutaneous coronary intervention of non-culprit vessels in a staged procedure during index admission.
  Arms: In-hospital complete revascularization group.
Other: After-discharge nonculprit-lesions percutaneous coronary intervention (PCI) — To perform percutaneous coronary intervention of non-culprit vessels in a staged procedure after hospital discharge.
  Arms: After-discharge complete revascularization group.

SUMMARY:
Patients with STEMI and multivessel disease in whom the culprit lesion has been successfully revascularized during prmimary PCI, will be randomized to in-hospital or after-discharge complete revascularization.

The purpose of this study is to evaluate the impact of these two different strategies in terms of hospital stay.

DETAILED DESCRIPTION:
STEMI patients with mutivessel disease are, after successful primary angioplasty, randomized 1:1 ratio to either in-hospital complete revascularization or after-discharge complete revascularization strategy.

Eligible non-culprit coronary arteries must be >2.0 mm in diameter and at the discretion of the operator suitable for PCI. Only arteries with angiographically stenoses ≥70% or between ≥50% and <70 in proximal segments can be randomized.

Patients in the in-hospital revascularization group will undergo to non-culprit percutaneous coronary intervention (PCI) at least 24 hours after ST-segment elevation myocardial infarction. On the other hand, patients in the after-discharge group will undergo to non-culprit PCI within 4-6 weeks after STEMI.

ELIGIBILITY:
Inclusion Criteria:

* Acute onset of chest pain <12 hours duration.
* ST-segment elevation ≥ 0.1 millivolt in ≥ 2 contiguous leads, signs of a true posterior infarction or documented newly developed left bundle branch block.
* Culprit lesion in a major native vessel, with successful primary PCI.
* Presence of at least one non-culprit lesion more than or equal to 70% of stenosis in a vessel more than 2mm of diameter or more than or equal to 50% stenosis in proximal segments.
* The patient is able to give written consent for participation in the study.

Exclusion Criteria:

* Pregnancy.
* Significant left main stenosis.
* Stent thrombosis.
* Chronic total occlusion.
* Severe stenosis of non-culprit vessels with distal flow less than TIMI3.
* Significant non-culprit stenosis no candidate to revascularization.
* Presence of valvulopathy candidate for cardiac surgery.
* Cardiogenic shock status at admission.
* The patient is not able to give written consent for participation in the study.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2018-01-20 (Actual); Primary Completion 2021-11-25 (Actual); Study Completion 2022-12-21 (Actual)

PRIMARY OUTCOMES:
Impact in hospital stay | 6 months
  To evaluate the impact of two different revascularization strategies (in-hospital versus after-discharge) in terms of hospital stay (days) in patients with a STEMI and multivessel disease.

SECONDARY OUTCOMES:
Cardiovascular death, acute myocardial infarction or revascularization. | 1 year
  Composite of cardiovascular death, myocardial infarction, or ischemia driven revascularization of non-culprit coronary lesions eligible for and randomized to either of the two strategies.
Fractional flow reserve of angiographically moderate stenosis | 6 months
  Evaluate the presence of ischemia by analyzing the fractional flow reserve of angiographically moderate stenoses (≥50% and <70) in proximal segments of the anterior descending, circumflex, or right coronary artery.

CONTACTS AND LOCATIONS:
Overall Officials: Eva Rumiz Gonzalez, MD, PhD, Principal Investigator — Hospital General Universitario de Valencia
Locations (1):
- Hospital General Universitario de Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Antman EM, Anbe DT, Armstrong PW, Bates ER, Green LA, Hand M, Hochman JS, Krumholz HM, Kushner FG, Lamas GA, Mullany CJ, Ornato JP, Pearle DL, Sloan MA, Smith SC Jr, Alpert JS, Anderson JL, Faxon DP, Fuster V, Gibbons RJ, Gregoratos G, Halperin JL, Hiratzka LF, Hunt SA, Jacobs AK, Ornato JP. ACC/AHA guidelines for the management of patients with ST-elevation myocardial infarction; A report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines (Committee to Revise the 1999 Guidelines for the Management of patients with acute myocardial infarction). J Am Coll Cardiol. 2004 Aug 4;44(3):E1-E211. doi: 10.1016/j.jacc.2004.07.014. No abstract available. PMID 15358047
- [Background] Keeley EC, Boura JA, Grines CL. Primary angioplasty versus intravenous thrombolytic therapy for acute myocardial infarction: a quantitative review of 23 randomised trials. Lancet. 2003 Jan 4;361(9351):13-20. doi: 10.1016/S0140-6736(03)12113-7. PMID 12517460
- [Background] Andersen HR, Nielsen TT, Vesterlund T, Grande P, Abildgaard U, Thayssen P, Pedersen F, Mortensen LS; DANAMI-2 Investigators. Danish multicenter randomized study on fibrinolytic therapy versus acute coronary angioplasty in acute myocardial infarction: rationale and design of the DANish trial in Acute Myocardial Infarction-2 (DANAMI-2). Am Heart J. 2003 Aug;146(2):234-41. doi: 10.1016/S0002-8703(03)00316-8. PMID 12891190
- [Background] O'Gara PT, Kushner FG, Ascheim DD, Casey DE Jr, Chung MK, de Lemos JA, Ettinger SM, Fang JC, Fesmire FM, Franklin BA, Granger CB, Krumholz HM, Linderbaum JA, Morrow DA, Newby LK, Ornato JP, Ou N, Radford MJ, Tamis-Holland JE, Tommaso CL, Tracy CM, Woo YJ, Zhao DX. 2013 ACCF/AHA guideline for the management of ST-elevation myocardial infarction: a report of the American College of Cardiology Foundation/American Heart Association Task Force on Practice Guidelines. J Am Coll Cardiol. 2013 Jan 29;61(4):e78-e140. doi: 10.1016/j.jacc.2012.11.019. Epub 2012 Dec 17. No abstract available. PMID 23256914
- [Background] Sorajja P, Gersh BJ, Cox DA, McLaughlin MG, Zimetbaum P, Costantini C, Stuckey T, Tcheng JE, Mehran R, Lansky AJ, Grines CL, Stone GW. Impact of multivessel disease on reperfusion success and clinical outcomes in patients undergoing primary percutaneous coronary intervention for acute myocardial infarction. Eur Heart J. 2007 Jul;28(14):1709-16. doi: 10.1093/eurheartj/ehm184. Epub 2007 Jun 7. PMID 17556348
- [Background] Hannan EL, Samadashvili Z, Walford G, Holmes DR Jr, Jacobs AK, Stamato NJ, Venditti FJ, Sharma S, King SB 3rd. Culprit vessel percutaneous coronary intervention versus multivessel and staged percutaneous coronary intervention for ST-segment elevation myocardial infarction patients with multivessel disease. JACC Cardiovasc Interv. 2010 Jan;3(1):22-31. doi: 10.1016/j.jcin.2009.10.017. PMID 20129564
- [Background] Vlaar PJ, Mahmoud KD, Holmes DR Jr, van Valkenhoef G, Hillege HL, van der Horst IC, Zijlstra F, de Smet BJ. Culprit vessel only versus multivessel and staged percutaneous coronary intervention for multivessel disease in patients presenting with ST-segment elevation myocardial infarction: a pairwise and network meta-analysis. J Am Coll Cardiol. 2011 Aug 9;58(7):692-703. doi: 10.1016/j.jacc.2011.03.046. PMID 21816304
- [Background] Wald DS, Morris JK, Wald NJ, Chase AJ, Edwards RJ, Hughes LO, Berry C, Oldroyd KG; PRAMI Investigators. Randomized trial of preventive angioplasty in myocardial infarction. N Engl J Med. 2013 Sep 19;369(12):1115-23. doi: 10.1056/NEJMoa1305520. Epub 2013 Sep 1. PMID 23991625
- [Background] Gershlick AH, Khan JN, Kelly DJ, Greenwood JP, Sasikaran T, Curzen N, Blackman DJ, Dalby M, Fairbrother KL, Banya W, Wang D, Flather M, Hetherington SL, Kelion AD, Talwar S, Gunning M, Hall R, Swanton H, McCann GP. Randomized trial of complete versus lesion-only revascularization in patients undergoing primary percutaneous coronary intervention for STEMI and multivessel disease: the CvLPRIT trial. J Am Coll Cardiol. 2015 Mar 17;65(10):963-72. doi: 10.1016/j.jacc.2014.12.038. PMID 25766941
- [Background] Engstrom T, Kelbaek H, Helqvist S, Hofsten DE, Klovgaard L, Holmvang L, Jorgensen E, Pedersen F, Saunamaki K, Clemmensen P, De Backer O, Ravkilde J, Tilsted HH, Villadsen AB, Aaroe J, Jensen SE, Raungaard B, Kober L; DANAMI-3-PRIMULTI Investigators. Complete revascularisation versus treatment of the culprit lesion only in patients with ST-segment elevation myocardial infarction and multivessel disease (DANAMI-3-PRIMULTI): an open-label, randomised controlled trial. Lancet. 2015 Aug 15;386(9994):665-71. doi: 10.1016/s0140-6736(15)60648-1. PMID 26347918
- [Background] Smits PC, Abdel-Wahab M, Neumann FJ, Boxma-de Klerk BM, Lunde K, Schotborgh CE, Piroth Z, Horak D, Wlodarczak A, Ong PJ, Hambrecht R, Angeras O, Richardt G, Omerovic E; Compare-Acute Investigators. Fractional Flow Reserve-Guided Multivessel Angioplasty in Myocardial Infarction. N Engl J Med. 2017 Mar 30;376(13):1234-1244. doi: 10.1056/NEJMoa1701067. Epub 2017 Mar 18. PMID 28317428
- [Background] Levine GN, Bates ER, Blankenship JC, Bailey SR, Bittl JA, Cercek B, Chambers CE, Ellis SG, Guyton RA, Hollenberg SM, Khot UN, Lange RA, Mauri L, Mehran R, Moussa ID, Mukherjee D, Ting HH, O'Gara PT, Kushner FG, Ascheim DD, Brindis RG, Casey DE Jr, Chung MK, de Lemos JA, Diercks DB, Fang JC, Franklin BA, Granger CB, Krumholz HM, Linderbaum JA, Morrow DA, Newby LK, Ornato JP, Ou N, Radford MJ, Tamis-Holland JE, Tommaso CL, Tracy CM, Woo YJ, Zhao DX. 2015 ACC/AHA/SCAI Focused Update on Primary Percutaneous Coronary Intervention for Patients With ST-Elevation Myocardial Infarction: An Update of the 2011 ACCF/AHA/SCAI Guideline for Percutaneous Coronary Intervention and the 2013 ACCF/AHA Guideline for the Management of ST-Elevation Myocardial Infarction. J Am Coll Cardiol. 2016 Mar 15;67(10):1235-1250. doi: 10.1016/j.jacc.2015.10.005. Epub 2015 Oct 21. No abstract available. PMID 26498666
- [Background] Ibanez B, James S, Agewall S, Antunes MJ, Bucciarelli-Ducci C, Bueno H, Caforio ALP, Crea F, Goudevenos JA, Halvorsen S, Hindricks G, Kastrati A, Lenzen MJ, Prescott E, Roffi M, Valgimigli M, Varenhorst C, Vranckx P, Widimsky P; ESC Scientific Document Group. 2017 ESC Guidelines for the management of acute myocardial infarction in patients presenting with ST-segment elevation: The Task Force for the management of acute myocardial infarction in patients presenting with ST-segment elevation of the European Society of Cardiology (ESC). Eur Heart J. 2018 Jan 7;39(2):119-177. doi: 10.1093/eurheartj/ehx393. No abstract available. PMID 28886621
- [Background] Politi L, Sgura F, Rossi R, Monopoli D, Guerri E, Leuzzi C, Bursi F, Sangiorgi GM, Modena MG. A randomised trial of target-vessel versus multi-vessel revascularisation in ST-elevation myocardial infarction: major adverse cardiac events during long-term follow-up. Heart. 2010 May;96(9):662-7. doi: 10.1136/hrt.2009.177162. Epub 2009 Sep 23. PMID 19778920
- [Background] Grines CL, Marsalese DL, Brodie B, Griffin J, Donohue B, Costantini CR, Balestrini C, Stone G, Wharton T, Esente P, Spain M, Moses J, Nobuyoshi M, Ayres M, Jones D, Mason D, Sachs D, Grines LL, O'Neill W. Safety and cost-effectiveness of early discharge after primary angioplasty in low risk patients with acute myocardial infarction. PAMI-II Investigators. Primary Angioplasty in Myocardial Infarction. J Am Coll Cardiol. 1998 Apr;31(5):967-72. doi: 10.1016/s0735-1097(98)00031-x. PMID 9561995
- [Derived] Rumiz E, Valero E, Fernandez C, Vilar JV, Pellicer M, Cubillos A, Berenguer A, Facila L, Vano J, Nunez J. In-hospital versus after-discharge complete revascularization in patients with ST segment elevation myocardial infarction and multivessel disease. REVIVA-ST trial. PLoS One. 2024 May 14;19(5):e0303284. doi: 10.1371/journal.pone.0303284. eCollection 2024. PMID 38743727